CLINICAL TRIAL: NCT06124794
Title: A Multicenter, Single Group, Open, Extension Study of Phase III Clinical Trial to Compare the Efficacy and Safety of Protoxin in Subjects With Moderate to Severe Glabellar Lines
Brief Title: The Efficacy and Safety of Protoxin in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protox Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT_BTA_P3_21_EXT
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-11

CONDITIONS: Glabellar Frown Lines
Keywords: Glabellar Lines; Botulinum toxin; Botulinum toxin type A

STUDY DESIGN:
Intervention Model Description: A Multicenter, Single group, Open, Extension Study of Phase III Clinical Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROTOXIN 100U (Clostridium botulinum toxin type A) (Experimental): PROTOXIN will be injected to 5 glabellar lines (Each 4U/0.1mL, Total 20U/0.5mL)
  Interventions: Biological: PROTOXIN

INTERVENTIONS:
Biological: PROTOXIN — Clostridium botulinum toxin type A

SUMMARY:
This clinical trial is an extended clinical trial for test subjects who participated in the phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number) and completed follow-up observation up to 16 weeks after administration of clinical trial drugs, and evaluates the effectiveness and safety of repeated administration of protoxin in those with moderate or severe brow wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* PT_BTA_P3_21 (clinical trial plan number) Test subjects who participated in clinical trials and completed follow-up observation up to 16 weeks after administration of clinical trial drugs
* Men and women aged between 19 to 65 years old
* Subjects attaining ≥grade 2(moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Those who understand and comply with clinical trial procedures and visit schedules
* Subjects who voluntarily decides to participate and signs the consent form after hearing the explanation of this clinical trial.

Exclusion Criteria:

1. A person who has or is accompanied by the following diseases at the time of screening

   1. A person with systemic neuromuscular junction disorder that can affect neuromuscular function [myasthenia gravis (MG), Lambert-Eaton myasthenic syndrome, amyotrophic lateral sclerosis (ALS), etc.]
   2. A person with a history of facial paralysis or ptosis
   3. A person who has skin abnormalities such as infections, skin diseases, scars, etc. at the site to be administered
2. A person who has wrinkles to the extent that the glabellar lines cannot be physically flattened, such as when wrinkles are not straightened by hand
3. A person who is taking the following drugs

   1. Within 4 weeks of screening: Drugs with muscle relaxation action, such as muscle relaxants, spectinomycin hydrochloride, aminoglycoside antibiotics, polypeptide antibiotics, tetracycline antibiotics, lincomycin antibiotics, anticholinergics, benzodiazepines and similar drugs, and benzamide drugs [However, for muscle relaxants, benzodiazepines and similar drugs, a person who has stably maintained administration of them from within 4 weeks from the time of screening (the same drug is maintained without changing the usage and dose), and is not expected to change in ingredients, usage, and dose of them during the clinical trial period can be enrolled]
   2. A person who has administered aspirin or NSAIDs within 7 days before administration of the investigational product (However, low-dose aspirin (100 mg/day or less) administered for antithrombotic purposes is permitted)
4. A person who has had procedure/surgery that may affect the wrinkles around the glabellar or forehead during the following period

   1. Within 48 weeks of screening: Tissue augmentation
   2. Within 24 weeks of screening: A person who has undergone facial plastic surgery including glabellar lines such as brow lift, dermal resurfacing, or peeling, etc.
5. A person with a history of surgery or treatment around the orbit (except for double eyelid surgery, epicanthal fold (Mongolian fold) correction)
6. A person who is planning to undergo facial cosmetic procedures such as dermal filler, photorejuvenation, chemical peeling, and dermabrasionduring the clinical trial period
7. PT_BTA_P3_21 (Clinical Trial Plan Number) A person who received similar drugs for clinical trials such as botulinum toxin A and B after visiting the end of phase 3 clinical trials)
8. A person who is expected to administer botulinum toxin formulations other than this investigational product during the clinical trial period
9. A person with a history of hypersensitivity or allergy to the components of the investigational product (botulinum toxin formulations and serum albumin, etc.)
10. A person with a history of alcohol or drug addiction
11. A person who, in the investigator's judgment, may affect clinical trial participation or objective efficacy evaluation results, due to anxiety disorders or other significant psychiatric disorders (e.g., severe depression)
12. Women and men of childbearing potential who plan to become pregnant or do not intend to use appropriate contraceptive methods* during the clinical trial period

    * Appropriate contraceptive methods
    1. Using either hormonal contraceptives (subcutaneous implants, injections, oral contraceptives, etc.) or spermicide in combination with physical barrier methods (condoms, contraceptive diaphragms, vaginal sponges, cervical caps)
    2. Implantation of an intrauterine device or intrauterine system: A copper loop, hormone-containing intrauterine system
    3. Both men (condoms) and women (contraceptive diaphragms, vaginal sponges or cervical caps) use physical barrier methods together
    4. Surgical sterilization procedure/surgery: Bilateral tubal ligation, vasectomy, etc.
13. Pregnant or lactating women
14. A person with serious comorbidities (e.g., malignant tumors, immunodeficiency (decreased immune function), renal disease, liver disease, heart disease, respiratory disease, etc.) or acute diseases that are unsuitable for participation in the clinical trial as judged by the investigator
15. A person who participated in other clinical trials/clinical device trials within 30 days prior to screening and received administration/treatment of investigational products/devices, or a person for whom the longer period has not passed between the above period and 5 times the half-life of the investigational product in the clinical trial in which they participated
16. Others who are judged inappropriate to participate in this clinical trial by the investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure : We will use FWS(Facial wrinkle scale) | 4 weeks post injection compared to baseline
  In the Phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number), the improvement rate of brow wrinkles at 4 weeks after the administration of protoxin week and the improvement rate at the time of raising at 4 weeks after the administration of protoxin week in this extended clinical trial are compared and evaluated.

SECONDARY OUTCOMES:
Secondary Outcome Measures : We will use FWS(Facial wrinkle scale) | Week 8, 12, 16
  In the Phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number), the improvement rate of brow wrinkles at 8, 12, and 16 weeks after the administration of protoxin week is compared with the improvement rate of brow wrinkles at 8, 12, and 16 weeks after the administration of protoxin week in this extended clinical trial.
Secondary Outcome Measures : We will use FWS(Facial wrinkle scale) | Week 4, 8, 12, 16
  In the Phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number), we compare the improvement rate of normal brow wrinkles according to the tester's field evaluation at 4, 8, 12, and 16 weeks after the protoxin injection with the usual brow wrinkles according to the tester's field evaluation at 4, 8, 12, and 16 weeks after the protoxin injection in this extended clinical trial.
Secondary Outcome Measures : We will use FWS(Facial wrinkle scale) | Week 4, 8, 12, 16
  In the Phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number), the improvement rate of normal brow wrinkles is compared with the improvement rate of normal brow wrinkles at 4, 8, 12, and 16 weeks after the administration of protoxin in this extended clinical trial.
Secondary Outcome Measures : We will use FWS(Facial wrinkle scale) | Week 4, 8, 12, 16
  In the phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number), the rate of improvement of brow wrinkles at 4, 8, 12, and 16 weeks after Botox week administration and the rate of improvement of brow wrinkles at 4, 8, 12, and 16 weeks after protoxin week administration in this extended clinical trial are compared and evaluated.
Secondary Outcome Measures : We will use FWS(Facial wrinkle scale) | Week 4, 8, 12, 16
  In the Phase 3 clinical trial of PT_BTA_P3_21 (clinical trial plan number), the proportion of test subjects satisfied in the satisfaction assessment of test subjects at 4, 8, 12, and 16 weeks after the administration of protoxin in this extended clinical trial is compared with the proportion of test subjects satisfied in the satisfaction assessment of test subjects at 4, 8, 12, and 16 weeks after the administration of protoxin.
Secondary Outcome Measures : We will use FWS(Facial wrinkle scale) | Week 4, 8, 12, 16
  In Phase 3 of PT_B, comparing the proportion of subjects satisfied in the satisfaction assessment of subjects at week 4, 8, 12, and 16 after the main administration of PT_P3_21 (clinical trial plan number), and the proportion of subjects satisfied in the satisfaction assessment of subjects at week 4, 8, 12, and 16 after the main administration of protoxin, in this extended clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Beomjoon Kim, PI, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Yangone Lee, CI, Principal Investigator — Konkuk University Medical Center; Jonghoon Lee, PI, Principal Investigator — Nown Eulji Medical Center
Locations (3):
- South Korea (3):
  - Chung-Ang University Hospital, Seoul, Gwangjin-gu
  - Konkuk University Hospital, Seoul, Gwangjin-gu
  - Nowon Eulji Medical Center, Seoul, Nowon-gu

IPD SHARING:
Plan to Share IPD: No